CLINICAL TRIAL: NCT03430492
Title: The Molecular Fingerprint of Psychological Resilience - Implications for Diagnostic and Therapeutic Strategies
Brief Title: Sweden Cancerome Analysis Network - Breast (SCAN-B) Coupled to Psychological Resilience
Status: Active, not recruiting | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Vinnova (Other Government); Mats Paulssons stiftelse, org. nr 802423-3150 (Unknown); Gunnar Nilsson's Cancer Foundation (Other); CREATE Health Cancer Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: SCAN-B Resilience
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Psychological Resilience; Biomarkers; Molecular Fingerprint; Quality of Life (QoL); Body and Mind; CD-RISC; SF-36
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to define the association between psychological resilience and biomolecular signatures in cancer patients and to relate psychological resilience to prognosis, as this could potentially open up a novel avenue of therapeutic interventions, medical as well as psychosocial.

DETAILED DESCRIPTION:
Individual patients differ in psychological response when receiving a cancer diagnosis. Given the same disease burden some patients master the situation well and others do experience a great deal of stress, depression and lowered quality of life. A patient's mental resistance after acquiring a threat, like a cancer diagnosis, called psychological resilience, is known to impact the outcome of the disease. Patients with high psychological resilience are likely to experience less stress reactions, and a better adaptation and management of the life threat and the demanding therapeutic interventions. How this phenomenon of mastering difficult situations is reflected also in bio-molecular processes is not much studied and how these have an impact on the cancer prognosis and the effectiveness of treatment is today not fully understood. However, there is evidence that expressing the emotions evoked is an important part of fighting cancer.

Our hypothesis is that patients displaying a high psychological resilience, according to a standardized method "The Connor-Davidson resilience scale" i.e. low stress reactions, low hopelessness and low fatigue, also present a specific pattern of biomolecular signatures in blood, represented by its epigenome, microRNA and proteomic patterns.

This project specifically aims to investigate if breast cancer patient´s psychological resilience can be coupled to bio-molecular parameters, using advanced "omics" and as a secondary aim, if it relates to prognosis and quality of life one year after diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with primary breast cancer
* Patients consented to be included in the SCAN-B study at (Blekinge County Hospital, Central Hospital Växjö and Hallands Hospital Halmstad HBG??
* Oral and written consent for the SCAN-B Resilience study
* Age ≥ 18 years
* Patients that do understand the Swedish language (written and spoken)

Exclusion Criteria:

* No diagnosis of breast cancer
* Not consented to be included in the SCAN-B study
* Do not understand the Swedish language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study includes only women with newly diagnosed breast cancer
Study Population: SCAN-B Resilience is, as a part of the SCAN-B program, a prospective breast cancer study with established infrastructure for enrollment and follow-ups for patient. The study population is newly diagnosed breast cancer patients enrolled in SCAN-B at the hospitals in Karlskrona, Helsingborg, Växjö and Halmstad.
  The INCA register (a information network for cancer care) includes almost 100% of all women diagnosed with breast cancer. Based on comparison with cancer registrations in INCA for 2011-2012, 85 % of all new breast cancer diagnosed women are included in SCAN-B. In April 2017 83% of patients included in SCAN-B were also enrolled in SCAN-B Resilience why a majority (70%) of women diagnosed with breast cancer are enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 985 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The association between psychological resilience and biomolecular signatures in breast cancer patients | All patients enrolled 2019-12-31. Analysis 2020-2022
  Measured by CD-RISC and bimolecular techniques.

SECONDARY OUTCOMES:
The association between psychological resilience and quality of life at baseline in breast cancer patients | All patients enrolled 2019-12-31. Analysis 2020-2022
  Measured by CD-RISC and SF-36
The association between psychological resilience and quality of life one year after diagnosis in breast cancer patients | Patients followed up one year from diagnosis. All patients enrolled 2019-12-31. Analysis 2020-2022
  Measured by CD-RISC and SF-36
The association between psychological resilience and recovery/rehabilitation five years after | Patients followed up five years from diagnosis. All patients enrolled 2019-12-31. Analysis 2020-2024
  Measured by CD-RISC and study specific questionnaire based on the Swedish national cancer rehabilitation guidelines.
The association between psychological resilience and prognosis in breast cancer patients | Patients followed up one year from diagnosis. All patients enrolled 2019-12-31. Analysis 2020-2024
  Measured by CD-RISC correlated to register data
The association between psychological resilience and clinicopathological characteristics | All patients enrolled 2019-12-31. Analysis 2020-2024
  Measured by CD-RISC and correlated to register data
The association between quality of life and clinicopathological characteristics | Patients followed one year from diagnosis. All patients enrolled 2019-12-31. Analysis 2020-2024
  Measured by SF-36 and correlated to register data

CONTACTS AND LOCATIONS:
Overall Officials: Carl AK Borrebaeck, Professor, Principal Investigator — Lund University
Locations (4):
- Sweden (4):
  - Blekinge County Hospital, Karlskrona, Blekinge County
  - Hallands Hospital Halmstad, Halmstad, Halland County
  - Helsingborgs hospital, Helsingborg, Skåne County
  - Central Hospital Växjö, Vaxjo, Småland

IPD SHARING:
Plan to Share IPD: Undecided
Upon publication, the relevant anonymized individual participant data will be shared.

REFERENCES:
- [Background] Saal LH, Vallon-Christersson J, Hakkinen J, Hegardt C, Grabau D, Winter C, Brueffer C, Tang MH, Reutersward C, Schulz R, Karlsson A, Ehinger A, Malina J, Manjer J, Malmberg M, Larsson C, Ryden L, Loman N, Borg A. The Sweden Cancerome Analysis Network - Breast (SCAN-B) Initiative: a large-scale multicenter infrastructure towards implementation of breast cancer genomic analyses in the clinical routine. Genome Med. 2015 Feb 2;7(1):20. doi: 10.1186/s13073-015-0131-9. eCollection 2015. PMID 25722745
- [Background] Axelsson U, Ryden L, Johnsson P, Eden P, Mansson J, Hallberg IR, Borrebaeck CAK. A multicenter study investigating the molecular fingerprint of psychological resilience in breast cancer patients: study protocol of the SCAN-B resilience study. BMC Cancer. 2018 Aug 6;18(1):789. doi: 10.1186/s12885-018-4669-y. PMID 30081937
- [Result] Mohlin A, Bendahl PO, Hegardt C, Richter C, Hallberg IR, Ryden L. Psychological Resilience and Health-Related Quality of Life in 418 Swedish Women with Primary Breast Cancer: Results from a Prospective Longitudinal Study. Cancers (Basel). 2021 May 6;13(9):2233. doi: 10.3390/cancers13092233. PMID 34066499
- [Result] Mohlin A, Axelsson U, Bendahl PO, Borrebaeck C, Hegardt C, Johnsson P, Rahm Hallberg I, Ryden L. Psychological Resilience and Health-Related Quality of Life in Swedish Women with Newly Diagnosed Breast Cancer. Cancer Manag Res. 2020 Nov 24;12:12041-12051. doi: 10.2147/CMAR.S268774. eCollection 2020. PMID 33269004
- [Result] Velickovic K, Borrebaeck CAK, Bendahl PO, Hegardt C, Johnsson P, Richter C, Ryden L, Hallberg IR. One-year recovery from breast cancer: Importance of tumor and treatment-related factors, resilience, and sociodemographic factors for health-related quality of life. Front Oncol. 2022 Aug 16;12:891850. doi: 10.3389/fonc.2022.891850. eCollection 2022. PMID 36052232
- See also: SCAN-B homepage — https://www.scan-b.lu.se